CLINICAL TRIAL: NCT03984513
Title: Surviving And Thriving In The Real World: A Daily Living Skills Intervention For Adolescents With ASD
Brief Title: Daily Living Skills Intervention for 9th and 10th Graders With Autism Spectrum Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIN-DUNCAN-2018-5606; 1K23HD094855-01A1 (NIH)
Record Dates: First submitted 2019-05-24; First posted 2019-06-13 (Actual); Results first posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial - A study in which the participants are divided by chance into separate groups that compare different treatments or other interventions.
Who Masked: Outcomes Assessor
Masking Description: Coordinator who is assessing goals of participants is masked from knowing which group each participant was randomized to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STRW (Experimental): Participants will receive the daily living skills intervention, Surviving and Thriving in the Real World (STRW).
  Interventions: Behavioral: Surviving and Thriving in the Real World
- PEERS (Active Comparator): Participants will receive a social skills intervention, Program for the Education and Enrichment of Relational Skills (PEERS).
  Interventions: Behavioral: Program for the Education and Enrichment of Relational Skills

INTERVENTIONS:
Behavioral: Surviving and Thriving in the Real World — The Surviving and Thriving in the Real World intervention consists of 14 weekly concurrent adolescent and parent group sessions. The daily living skills to be targeted in the intervention include: Morning Routine (i.e., completing a morning personal hygiene routine); Laundry (i.e., sorting clothing, using a washing machine and dryer, and folding and putting clothes away); Kitchen/Cooking (i.e., cooking items in the microwave, oven, and stove, safe kitchen practices, cleaning up the kitchen after cooking, and grocery shopping); Self-Management (i.e., managing worry and stress related to learning daily living skills and transitioning to adulthood); and Money Management (i.e., using money to purchase items, evaluating the quality and price of items, understanding and using a checking and savings account, and budgeting money to cover expenses).
  Arms: STRW
Behavioral: Program for the Education and Enrichment of Relational Skills — Program for the Education and Enrichment of Relational Skills is an evidence-based social skills training program for youth with social challenges between the ages of 13-18.The program includes a teen group and a parent group that meet concurrently. Teens learn about conversations, electronic communication, joining groups, humor, handling teasing and disagreements, and planning a get-together with other teens. Parents learn how to coach their teens to continue to use the skills when the program is complete.
  Arms: PEERS

SUMMARY:
The current study seeks to develop the first daily living skills (DLS) intervention package for high functioning adolescents with autism spectrum disorder (ASD) and evaluate its effectiveness. The investigators hope to further refine the Surviving and Thriving in the Real World (STRW) intervention by conducting an ORBIT (Obesity-Related Behavioral Intervention Trial) Phase 2b feasibility Randomized Clinical Trial (RCT). This randomized clinical trial will test the preliminary effectiveness of STRW in 56 adolescents (14-21 years) with high functioning ASD as compared to a robust evidence-based social skills intervention (Program for the Evaluation and Enrichment of Relational Skills - PEERS). The current proposal represents a critical step toward improving the adult outcome of individuals with autism.

DETAILED DESCRIPTION:
Individuals with high functioning autism are not developing the skills necessary to successfully transition from adolescence to college, employment, and independent living. Daily living skills (DLS) have been linked to positive adult outcome in individuals with autism. Studies have consistently found that adults with high functioning autism who have better developed daily living skills were more likely to attend college, be employed, have more meaningful social relationships, and have an increased quality of life as compared to those with poor daily living skills. A complex set of environmental, individual, and family factors likely affect the ability of adolescents with high functioning autism to acquire critical daily living skills. There are currently no evidence-based daily living skills intervention packages for adolescents with high functioning autism that would prepare them for independence in adulthood.

The current study involving human subjects consists of (1) a measurement development phase to develop, adapt, and pilot objective outcome measures of daily living skills and (2) a feasibility randomized clinical trial to test the feasibility and effectiveness of the Surviving and Thriving in the Real World intervention as compared to a social skills intervention. For the measurement development phase, 2 outcome measures (i.e., Daily Phone Diaries (DPDs) and behavioral observation measures of targeted daily living skills) will be developed/adapted and piloted with approximately 10 adolescents with autism between the ages of 14-21 and their parents. For the feasibility randomized clinical trial to test the preliminary effectiveness of Surviving and Thriving in the Real World, a total of 56 adolescents with autism between the ages of 14-21 will be randomized to Surviving and Thriving in the Real World (n=28) or a social skills group (n=28). Outcome measures will be assessed at baseline, post-treatment, and 6-month follow-up.

Power Analyses: The feasibility randomized clinical trial is being conducted with the intent of examining the differences in daily living skills to be expected. Few studies have examined the trajectory of daily living skills in individuals with autism, and no studies have examined how daily living skills develop during adolescence. Power calculations focused on the anticipated increase or improvement in the age equivalence scores of each of the Vineland-3 daily living skills subdomains for the Surviving and Thriving in the Real World group and control group. The investigators used conservative estimates of change in daily living skills subdomain age equivalence scores for the investigator's sample size estimation, even though a recent pre-post trial and pilot randomized clinical trial on Surviving and Thriving in the Real World found a mean improvement of 2.3 to 2.6 years across the 3 subdomains from baseline to post-treatment.

Aim 1: For each Vineland-3 daily living skills subdomain, the investigators anticipate that adolescents in the Surviving and Thriving in the Real World group will have a mean improvement of 11 months (a mean gain in age equivalence of 11 months) at post-treatment compared to a mean improvement of 4 months in the control group. Assuming a conservative pooled standard deviation of 8.4, the investigators will have 80% power to detect the above effect size (of 0.8) with 24 participants per group. Accounting for a potential 15% drop out rate, the effective sample size is 28 per group. Based on the investigator's past studies, the investigators would expect the mean improvement in the Surviving and Thriving in the Real World group to be 16 months, but the investigators wanted to be conservative and estimate the sample size based on detecting a mean improvement as small as 11 months in the Surviving and Thriving in the Real World group.

Aim 2: For each daily living skills subdomain, the investigators anticipate that all participants who receive the Surviving and Thriving in the Real World treatment will maintain treatment gains from post-treatment to 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* attending high school
* a diagnosis of autism spectrum disorder (ASD) (based on meeting the cut-off score on the Autism Diagnostic Observation Schedule, 2nd Edition.
* a full scale Intelligence Quotient (IQ) of 70 or above as measured by the Stanford Binet Intelligence Scales, 5th Edition.
* deficient daily living skills as assessed by the Vineland-3.

Exclusion Criteria:

* psychosis or other major psychiatric disorder requiring intensive treatment
* the adolescent has already completed the social skills group (PEERS), either at Cincinnati Children's or in another setting, unless it has been a significant amount of time since they did the PEERS group (2-3 years, or up to the discretion of the PI).

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amie M Duncan, Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited using flyers via our hospital's outpatient autism clinic, research databases, and within the community.
Pre-assignment Details: We had several screen fails, which we compensated for by enrolling above our target number for completion.
Period: Overall Study
Arm/Group | STRW | PEERS
Started | 29 | 29
Completed | 26 | 22
Not Completed | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | STRW | PEERS | Total
Number analyzed (Participants) | 26 | 22 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26 | 22 | 48
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 10 | 13
  Male | 23 | 12 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 23 | 17 | 40
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 22 | 48
Vineland-3 Baseline DLS Domain Standard Score [Mean (Standard Deviation); unit: units on a scale] — A measure of adaptive behavior that assesses skills in the Communication, Daily Living Skills, and Socialization domains. The Daily Living Skills domain is comprised of the Personal, Domestic, and Community subdomains and has items that directly correspond to goals being targeted in the current study.
  The range of standard scores for the Daily Living Skills domain is 20 to 140. Standard scores have a mean of 100 and a standard deviation of 15. A higher standard score indicates a higher level of adaptive behavior.
  units on a scale | 64.0 (13.6) | 54.8 (22.5) | 59.4 (18.05)

OUTCOME MEASURES:

1. Primary Outcome: Vineland Adaptive Behavior Scales, 3rd Edition
Description: The Vineland Adaptive Behavior Scales, 3rd Edition (VABS-3) is a well-established standardized measure of adaptive behavior that assesses skills in the Communication, Daily Living Skills, and Socialization domains. The DLS domain is comprised of the Personal, Domestic, and Community subdomains and has items that directly correspond to goals being targeted in the STRW intervention.
  If you add the total points possible for each subdomain, the total Daily Living Skills Domain raw scores can range from 0 to 286. The higher the score, the better the adaptive level.
Time Frame: At Baseline, at Post-Group (approx. 3 months)
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | STRW | PEERS
Number analyzed (Participants) | 26 | 22
Score on a scale
  Daily Living Skill Domain Raw Score at Baseline | 199.0 (6.1) | 177.9 (5.4)
  Daily Living Skill Domain Raw Score at Post Group | 228.8 (7.1) | 203.3 (6.4)

ADVERSE EVENTS:
Time Frame: Each participant completed 3 visits and a group intervention over the course of about a 12 month period.
Arm/Group | STRW | PEERS
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/22
Other Adverse Events (participants affected / at risk) | 0/26 | 0/22

LIMITATIONS AND CAVEATS:
Limitations of the current study include use of a caregiver report measure for the primary outcome, a relatively small sample size, and the need for a more diverse sample of autistic teens.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-02): https://cdn.clinicaltrials.gov/large-docs/13/NCT03984513/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT03984513/ICF_001.pdf